CLINICAL TRIAL: NCT04399213
Title: Dermal Blood Flow Response to Escalating Doses of Histamine, Administered by a Skin Prick
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CCP18-3305-HIS-Part I
Record Dates: First submitted 2018-11-08; First posted 2020-05-22 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — Histamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): From cubital fossae to wrist: 50 - 15 - 5 µg histamine dihydrochloride
  Interventions: Procedure: 50 µg Histamine; Procedure: 15 µg Histamine; Procedure: 5 µg Histamine; Procedure: Placebo (saline)
- Group B (Experimental): From cubital fossae to wrist: 15 - 5 - 50 µg histamine dihydrochloride
  Interventions: Procedure: 50 µg Histamine; Procedure: 15 µg Histamine; Procedure: 5 µg Histamine; Procedure: Placebo (saline)
- Group C (Experimental): From cubital fossae to wrist: 5 - 50 - 15 µg histamine dihydrochloride
  Interventions: Procedure: 50 µg Histamine; Procedure: 15 µg Histamine; Procedure: 5 µg Histamine; Procedure: Placebo (saline)

INTERVENTIONS:
Procedure: 50 µg Histamine — Skin prick through 50 µg/5 µL histamine diHCl
Procedure: 15 µg Histamine — Skin prick through 15 µg/5 µL histamine diHCl
Procedure: 5 µg Histamine — Skin prick through 5 µg/5 µL histamine diHCl
Procedure: Placebo (saline) — Skin prick through 5 µL saline (0.9% NaCl)

SUMMARY:
To determine the effective dose and the time course, the dermal blood flow response to histamine will be evaluated at different doses (5 µg, 15 µg and 50 µg). Histamine will be administered by a skin prick on the volar surface of subjects' forearm, alongside a negative control. Changes in dermal blood flow will be measured with laser Doppler imaging at different time points following the skin prick.

ELIGIBILITY:
Inclusion criteria:

* Subject is a white male ≥ 18 and ≤ 45 years of age at the time of screening
* Subject is a nonsmoker for at least 6 months prior to the study start
* Subject has a body mass index ≥ 18 and ≤ 30 kg/m2
* Subject is judged to be in good health on the basis of medical history, physical examination and vital signs
* Subject understands the procedures and agrees to comply with them for the entire length of the study by giving written informed consent

Exclusion criteria:

* Subject has excessive hair growth on the volar surface of the forearm
* Subject has a past or present history of diffuse dermatological conditions including eczema, scleroderma, psoriasis, urticaria, dermatographism and dermatitis
* Subject has any abnormality on the skin of the forearm, possibly interfering with the study assessments including tattoos, keloids, tumors, ulcers, burns, flaps and grafts
* Subject cannot avoid excessive tanning (any exposure to sunlight or a tanning bed which would cause a sunburn reaction) throughout the study and cannot cover the forearms 24 hours before and after each study visit
* Subject currently uses lotions, oils, depilatory preparations, makeup or other topical treatments on the arms and on a regular basis which cannot be discontinued for the duration of the study; subject has used any topical treatments within 7 days of the start of the study
* Subject has a past or present history of (symptomatic) asthma
* Subject has a history of severe allergic reactions to food or drugs or adverse experiences of a serious nature related to the administration of either a marketed or investigational drug, including histamine
* Subject currently uses any prescription or nonprescription drugs on a regular basis which cannot be discontinued for the duration of the study; subject has used any prescription or nonprescription medication within 14 days of the start of the study
* Subject is a habitual and heavy consumer of coffee or caffeinated beverages (more than approximately 4 cups of tea, coffee or cola per day) at the time of the study. Subjects who have reduced their consumption to ≤ 4 cups per day at least 1 week prior to enrollment may participate. Subjects who cannot refrain from caffeinated beverages 24 hours before the study visit
* Subject is unable to refrain from drinking alcohol 24 hours prior to histamine application, is currently a regular user (including "recreational use") of any illicit drugs, or has a history of drug (including alcohol) abuse. A drug screen will include amphetamines/ methamphetamines, methylenedioxymethamphetamine, benzodiazepines, barbiturates, cocaine, cannabis, tricyclic antidepressants, methadone and opiates
* Subject cannot refrain from being around second hand smoke 24 hours prior to histamine application or uses nicotine-containing products. Ex-smokers should have ceased smoking at least 6 months prior to screening
* Subject has any of the following vital sign measurements at screening: heart rate ≤ 40 or ≥ 100 beats/min, diastolic blood pressure ≤ 50 or ≥ 89 mmHg and/or systolic Blood Pressure ≤ 90 or ≥ 139 mmHg
* Subject has been involved in testing an investigational drug in another clinical study within the last 4 weeks or 5 half-lives
* Subject has evidence of a clinically significant active infection, fever of 38°C or above at the time of the study visits
* Subject has a history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs
* Subject is in a situation or has a condition, which, in the opinion of the investigator, may interfere with safe and optimal participation in the study
* Subject has a history of any illness or disorder, which, in the opinion of the investigator, might confound the results of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Change in dermal blood flow induced by histamine skin pricks, compared to baseline and placebo for different doses | The dermal blood flow will be assessed before (baseline) and every 5 minutes during the hour following the skin pricks

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Pharmacology, Leuven, Belgium